CLINICAL TRIAL: NCT03255746
Title: HELP-HY: Health Education and sLeep Program in HYpertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-004044; R01HL134808 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-08-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prehypertension; Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Enhancement (Experimental)
  Interventions: Behavioral: Sleep Enhancement
- Health Education (Placebo Comparator)
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Sleep Enhancement — This regimen combines education and behavioral skills to enable prolonging sleep in chronically sleep deprived subjects so as to better meet participant's sleep needs. This intervention emphasizes plain language communication of cognitive behavioral therapy strategies for initiating and maintaining health behavior change, primarily through using brief action plans (time-limited, personally relevant, behavioral goal setting with confidence), and collaborative problem-solving. Coaching will be provided to modify daily routines and adhere to sleep hygiene practices to allow for extended time in bed.
  Arms: Sleep Enhancement
Behavioral: Health Education — This is a placebo/attention control condition. Participants will receive health education based on NIH information. Number, duration, and frequency of sessions will be identical to those administered to the intervention group.
  Arms: Health Education

SUMMARY:
Hypertension is the major risk factor for cardiovascular and cerebrovascular diseases worldwide. The escalating prevalence of inadequate sleep now parallels that of hypertension. Observational and experimental evidence favoring a causal relation between insufficient sleep and hypertension are particularly compelling - sleeping 6 hours or less per night is associated with a 20-32% higher probability of incident hypertension. Since sleep curtailment is largely voluntary, sleep deficiency may be corrected and the detrimental health consequences potentially reversed.

In this study the investigators aim to investigate the effects of 8 weeks of sleep enhancement/extension vs health education in prehypertensive and stage 1 hypertensive subjects who report habitual short sleep (≤6.5 hours/night).

ELIGIBILITY:
Inclusion criteria:

* Age: 18 to 65 (inclusive)
* Gender: both males and females
* Body mass index (BMI): 18.5-34.9 kg/m2
* Habitual sleep duration <7 hours and voluntary prolongation of sleep when circumstances allow (as indicated by napping and/or >45 min catch-up sleep during weekends or holidays)
* Presence of prehypertension (office systolic BP (SBP) 120-139 mmHg and/or diastolic BP (DBP) 80-89 mmHg) , Stage 1 hypertension (office SBP 140-159 mmHg and/or DBP 90-99 mmHg ) , or currently taking antihypertensive medications
* Either on no prescription medications (other than oral contraceptive pills, or intrauterine devices) or on stable medical regimen for at least 1 month, if taking prescription medications for chronic conditions
* Not pregnant or breast feeding and not intending to become pregnant or breast feed
* Not a current smoker or tobacco user
* Ability to provide written informed consent.

Exclusion criteria:

* Vulnerable study populations will be excluded
* Pregnancy
* Smoking
* Shift-work
* Travel across >2 time zones in the previous month
* Presence of overt cardiovascular diseases, diabetes, chronic kidney disease, cancer, sleep/circadian disorders, psychiatric disorders
* If taking prescription medications for chronic conditions, change in therapy (type, frequency and/or dosage) over the previous month
* Sleep aids
* Habitual sleep duration ≥7 hours
* Excessive alcohol (>14 drinks/week in men and >7 drinks/week in women) and/or excessive caffeine intake (>400 mg)
* Currently on a diet and/or actively trying to lose weight
* History of drowsing driving
* Severe daytime sleepiness (score >15 at the Epworth Sleepiness Scale)
* Current or previous (during the past 2 months) participation in other research studies at the discretion of study personnel
* Blood/plasma donation during the past 2 months
* Unwillingness or inability to adjust sleep schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
change in 48-hour mean arterial pressure | 8 weeks
  changes in ambulatory measure of blood pressure

SECONDARY OUTCOMES:
changes in 48-hour heart rate | 8 weeks
  changes in 24-hour heart rate
changes in baroreflex sensitivity | 8 weeks
  changes in baroreflex sensitivity
changes in endothelial function | 8 weeks
  changes in endothelial function
changes in renin | 8 weeks
  changes in renin
changes in angiotensin peptides | 8 weeks
  changes in angiotensin peptides
changes in aldosterone | 8 weeks
  changes in aldosterone
changes in insulin sensitivity | 8 weeks
  changes in insulin sensitivity
changes in cortisol | 8 weeks
  changes in cortisol
changes in body fat | 8 weeks
  changes in body fat
changes in catecholamines | 8 weeks
  changes in catecholamines

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No